CLINICAL TRIAL: NCT02733666
Title: Open Reduction and Internal Fixation of Lateral Humeral Condyle Fractures With Absorbable Screws in Children
Brief Title: Internal Fixation of Lateral Humeral Condyle Fractures With Absorbable Screws in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuxi Su, Vice chief of the orthopeadic department of Children's Hospital of Chongqing Medical Univeristy, Children's Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yuxi-2016-3-25
Record Dates: First submitted 2016-03-25; First posted 2016-04-11 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Humeral Fractures
Keywords: Absorbable screw; Internal fixation; Children
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorbable screw group (Experimental): One absorbable screw was used for fixation in the experimental group
  Interventions: Procedure: Absorbable screw group
- K-wires group (No Intervention): two 1.8-mm K-wires were used for the fixation in the control group. The K-wires were the most common used by the orthopaedic surgeon.

INTERVENTIONS:
Procedure: Absorbable screw group — Open reduction was performed and one absorbable screw was used for fixation in the experimental group
  Arms: Absorbable screw group

SUMMARY:
Lateral humeral condyle fractures are the second most common elbow fractures in children. Displaced and rotated fractures require stabilization and reduction. Kirschner wires (K-wires) are most commonly used for fracture fixation. Here, the investigators introduce a new fixation method involving absorbable screws. The investigators aimed to determine if it is feasible to treat lateral humeral condyle fractures with absorbable screws by comparing the functional outcomes obtained using screw fixation vs. K-wire fixation.

DETAILED DESCRIPTION:
Methods: Between May 2007 and September 2010, 86 participants (age, 1.6-13 years; average age, 6.7 years) were randomly divided into two groups. All participants had been diagnosed with lateral condyle fractures classified as Jacobs type II (unstable) or III. Closed reduction failed in all participants. Therefore, open reduction was performed under general anesthesia. One absorbable screw was used for fixation in the experimental group, while two 1.8-mm K-wires were used in the control group. At 4-6 weeks postoperatively, the participants' plaster casts were removed, and functional training was started.

ELIGIBILITY:
Inclusion Criteria:

All participants had been diagnosed with lateral condyle fractures classified as Jacobs type II (unstable) or III

Exclusion Criteria:

participants had not been diagnosed with lateral condyle fractures classified as Jacobs type II (unstable) or III

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2007-05; Primary Completion 2010-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Elbow Motion angle in degree | 6 months after surgery.
  The orginal position was anatomy position （neutral position），Then，test the angle measured in degree of the elbow motion flexion, pronation and supination
Strength in Newton (N) | 6 months after surgery.
  Compared to the normal hand, the investigators defined it normal to moderate loss and severe loss
stability | 6 months after surgery.
  Compared to the normal hand, the investigators defined the elbow stability from normal to mild loss , moderate loss and severe loss
Pain | 6 months after surgery.
  According to the level 0 ~ 10 to pain grading:0 to 3 for mild pain,4 to 6 for moderate pain,7 or more for severe pain

IPD SHARING:
Plan to Share IPD: Undecided